CLINICAL TRIAL: NCT00844623
Title: Phase I Clinical Trial Of Gene Therapy For Hepatocellular Carcinoma By Intratumoral Injection Of TK99UN (An Adenoviral Vector Containing The Thymidine Kinase Of Herpes Simplex Virus)
Brief Title: TK-based Suicide Gene Therapy for Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Principal Investigator, Bruno Sangro Gomez-Acebo, Main investigator, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TK99UN-HCC1
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Carcinoma, Hepatocellular
Keywords: primary liver cancer, hepatoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: TK99UN — escalated dosis from 2x10e10 to 2x10e12 viral particles injected intratumorally
  Other Names: Adenoviral vector encoding for HSV-TK

SUMMARY:
The purpose of this study is to determine whether activation of a prodrug after intratumoral gene transfer is safe in humans, and to determine dose levels for further clinical development.

DETAILED DESCRIPTION:
The study is a phase I clinical trial evaluating the intratumoral injection of defective adenovirus containing HSVtk (the thymidine kinase of herpes simplex virus), in patients with advanced hepatocellular carcinoma that were not amenable to curative therapy. The study was conducted in a single center in Spain. Five consecutive cohorts of two patients received increasing doses of the vector by intratumoral injection and equal doses of either intravenous ganciclovir or oral valganciclovir. The dose received by each consecutive cohort of patients was progressively higher according to a prefixed scale.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal diagnosis of hepatocellular carcinoma according to histological confirmation or EASL-AASLD criteria
* Contraindication for surgical treatment of the disease
* Detectable disease by imaging
* Ability to give informed consent and to express the willingness to fulfill protocol requirements during the study

Exclusion Criteria:

* Current pregnancy or breast-feeding
* Acute infection
* Positive anti-HIV antibodies
* Hematologic alterations not attributable to hypersplenism, or in any case, intense neutropenia and thrombocytopenia, defined as neutrophil count lower than 0,5/pL or platelet count lower than 20/pL
* Participation in other clinical trial during the previous month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-12; Primary Completion 2003-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Daily for the first 16 day, monthly thereafter for 6 months, 3-monthly since then

SECONDARY OUTCOMES:
Tumor response by WHO criteria | at day 63 and months 4, 6, 9 y 12

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Prieto, MD, Principal Investigator — Clinica Universitaria de Navarra; Bruno Sangro, MD, Study Director — Clinica Universitaria de Navarra
Locations (1):
- Clinica Universitaria de Navarra, Pamplona, Spain

REFERENCES:
- [Background] Penuelas I, Mazzolini G, Boan JF, Sangro B, Marti-Climent J, Ruiz M, Ruiz J, Satyamurthy N, Qian C, Barrio JR, Phelps ME, Richter JA, Gambhir SS, Prieto J. Positron emission tomography imaging of adenoviral-mediated transgene expression in liver cancer patients. Gastroenterology. 2005 Jun;128(7):1787-95. doi: 10.1053/j.gastro.2005.03.024. PMID 15940613
- [Result] Sangro B, Mazzolini G, Ruiz M, Ruiz J, Quiroga J, Herrero I, Qian C, Benito A, Larrache J, Olague C, Boan J, Penuelas I, Sadaba B, Prieto J. A phase I clinical trial of thymidine kinase-based gene therapy in advanced hepatocellular carcinoma. Cancer Gene Ther. 2010 Dec;17(12):837-43. doi: 10.1038/cgt.2010.40. Epub 2010 Aug 6. PMID 20689572